CLINICAL TRIAL: NCT05882500
Title: Osteopontin and Other Potential Biomarkers and Factors Important for Prognosis in Pancreatitis
Brief Title: Osteopontin as a Biomarker in Pancreatitis
Acronym: PtitStudien
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Bergthor Björnsson, Associate Professor, Linkoeping University
Other Study IDs: PtitStudien
Record Dates: First submitted 2023-05-11; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreatits: Patients with pancreatitis based ont the Atlanta criteria
  Interventions: Other: No intervention, observation

INTERVENTIONS:
Other: No intervention, observation

SUMMARY:
In the early phase of pancreatits, factors that can give information about the development of severety are still lacking. In this study patients will be included prospectively upon the diagnosis of pancreatits and clinical as well as labarotory and radiological factors will be sampled. The aim is do identifiy factors that may aid in the risk stratification for development of different severity grades of pancreatitis.

DETAILED DESCRIPTION:
In the early phase of pancreatits, factors that can give information about the development of severety are still lacking. In this study patients will be included prospectively upon the diagnosis of pancreatits and clinical as well as labarotory and radiological factors will be sampled. The aim is do identifiy factors that may aid in the risk stratification for development of different severity grades of pancreatitis.

Patients admitted and diagnosed with pancreatitis (according to the Atlanta criteria) will have serial testing of se-osteopontin in addiation to rutine blood work. Computet tomograpy and chest x-ray are mandatory as is blood culture.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pancreatitis

Exclusion Criteria:

* Pregnancy, lactation, unable to understand the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2011-03-03 (Actual); Primary Completion 2016-10-19 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Se-osteopontin | Within 3 days from diagnosis
  Se-osteopontin will be measured at admission and on day 2 and 3 of hospital stay. The change over time will be correlated to severety of pancreatitis as classified in the current Atlanta classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Linkoping University Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No